CLINICAL TRIAL: NCT03094728
Title: Role of Human Leukocyte Antigen Matching in Liver Transplantation and Its Relation to Outcomes
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Fawzy Montasser, Clinical professor, Ain Shams University
Other Study IDs: HLA and liver transplantation
Record Dates: First submitted 2017-03-18; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver transplantation receipients: All patients underwent Living donor liver transplantation at Ain Shams center for organ transplantation (ASCOT) during the designed study period
  Interventions: Diagnostic Test: HLA cross matching

INTERVENTIONS:
Diagnostic Test: HLA cross matching — HLA Typing and Mismatch
  Cross matching (total and autocross):
  Cross match involves placing recipient serum onto donor lymphocytes and a cytotoxic reaction (deemed 'positive') suggests the presence of preformed donor specific antibodies (DSAs),Second, the original crossmatch should be repeated with the addition of the agent Dithiothreitol (DTT). DTT reduces the disulfide bonds in IgM thereby preventing IgM antibodies from generating a positive result.

SUMMARY:
The study aimed to assess HLA compatibility, HLA antibodies and cross matching in liver transplantation recipients and their relation to acute rejection, CMV infection, and recurrence of HCV.

DETAILED DESCRIPTION:
This was a cohort study conducted in patients who had undergone LDLT between January 2015 and January 2016 at in Ain Shams Center for Organ Transplantation (ASCOT) .

HLA Typing and Mismatch:

Preoperative blood samples from all recipients and donors were collected. The serological tissue typing for HLA was performed by a SSP-PCR (sequence-specific- primer). HLA-A, HLA- B, and HLA-DR loci were examined and used to calculate mismatch scores. The locus-specific type of HLA mismatch, as well as the degree of HLA mismatch, was then assessed. For each locus individually, the mismatch number was scored as 0, 1, or 2, on the basis of the number of donor alleles not shared with the respective recipient. Each patient was assigned an overall total score depending on the total number of mismatches at the 3 loci, ranging from 0 (no mismatches at any loci) to 6 (mismatches at all loci)

Cross matching (total and autocross):

Crossmatch involves placing recipient serum (potentially containing donor-specific anti-HLA antibodies) onto donor lymphocytes (containing HLA antigens).A cytotoxic reaction (deemed 'positive') suggests the presence of preformed DSAbs (donor specific antibodies).

Autoantibodies are generally IgM rather than IgG antibodies. To establish if autoantibodies are responsible for the result an auto-crossmatch should be performed. In this assay, recipient serum is crossmatched against recipient (rather than donor) lymphocytes. Second, the original crossmatch should be repeated with the addition of the agent Dithiothreitol (DTT). DTT reduces the disulfide bonds in IgM thereby preventing IgM antibodies from generating a positive result. IgM antibodies are generally regarded as having no pathological significance in transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Recipient selection:

  1. Adult recipients who are candidate for LDLT due to HCV related ESLD and meeting the transplantation criteria of the Ain Shams Center of Organ Transplantation (Child Pugh score ≥ 7and MELD score ≥15).

Donor selection:

1. Living donors are usually close family members or spouses, although unrelated living donors can be accepted according to the legal registration of MOH (ministry of health)
2. ABO blood type compatibility
3. Age is between 18-50
4. Absence of previous significant abdominal surgery and/or medical problems

Exclusion Criteria:

* Adult recipients who underwent LDLT due to other causes rather than HCV.
* Cardiopulmonary disease that cannot be corrected and is a prohibitive risk for surgery
* Acquired immunodeficiency syndrome (AIDS)
* Malignancy outside of the liver not meeting oncologic criteria for cure
* Hepatocellular carcinoma with metastatic spread
* Anatomic abnormalities that preclude liver transplantation
* Uncontrolled sepsis
* Acute liver failure with a sustained intracranial pressure >50 mmHg or a cerebral perfusion pressure <40 mmH
* Persistent non adherence with medical care and Lack of adequate social support
* Advanced age older than 65y.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with end stage liver diseases potential candidates for living donor liver transplantation and their donors
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Relation between HLA cross matching and post transplantation outcome | 1 year
  We o investigated the post transplantation laboratory data, incidence of acute rejection, recurrence of hepatitis C virus (HCV) infection and CMV infection as outcome parameters.

IPD SHARING:
Plan to Share IPD: Undecided